CLINICAL TRIAL: NCT00579787
Title: A Prospective Study Assessing the Emotional, Sexual and Quality of Life Concerns Of Women Undergoing Radical Trachelectomy Versus Radical Hysterectomy For Treatment Of Early Stage Cervical Cancer
Brief Title: Prospective Study Assessing Emotional, Sexual and Quality of Life Concerns Of Women Undergoing Removal of the Cervix Versus Removal of the Uterus,Ovaries and Fallopian Tubes For Treatment Of Early Stage Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Jeanne Carter, PhD, Memorial Sloan Kettering Cancer Center
Other Study IDs: 03-148
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; quality of life assessment; behavioral
MeSH Terms: conditions — Uterine Cervical Neoplasms; Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Women with early stage cervical cancer undergoing radical trachelectomy
- 2: Women with early stage cervical cancer undergoing radical hysterectomy

SUMMARY:
The purpose of this study is to will help us understand how two treatments impact women with early stage cervical cancer: a radical hysterectomy, which removes the entire uterus, the ovaries, and fallopian tubes versus a radical trachelectomy which removes the cervix, which is the bottom part of the uterus. The second leaves the rest of the uterus, the ovaries, and fallopian tubes. This means that there is a chance that the woman might be able to get pregnant in the future with this type of treatment. We believe that these two operations need further study to see how they impact women. This study will look at emotions and issues of fertility. The study will also ask about quality of life and sexual functioning. What we learn from this study will help us give better information to women considering these treatments.

DETAILED DESCRIPTION:
This project will prospectively assess and describe the emotional, sexual and quality of life impact of radical trachelectomy in comparison to the standard treatment of radical hysterectomy in women with early stage cervical cancer over a two year time period. Women being considered for radical trachelectomy with laparoscopic pelvic lymphadenectomy or radical hysterectomy (abdominal, laparoscopic or schauta) will be approached for study participation prior to undergoing surgery. After providing informed consent, participants will be given a survey questionnaire pre-operatively and asked to complete follow-up surveys post-operatively at follow up medical appointments at 3 months, 6 months, 12 months, 18 months and 24 months. We will assess the following domains in these women; mood, sexual functioning, and quality of life in addition to issues of fertility and treatment choice. The survey will take approximately 30 minutes to complete. The findings will be used to provide additional information to women considering these procedures and enable future interventions to be designed to meet any identified needs. In addition, the findings of this study will also be presented for consideration of a multi-center feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be suitable surgical candidates and completed the surgical consenting process with their gynecologic oncology surgeon.
* Confirmed invasive cervical cancer: squamous, adeno, or adenosquamous.
* FIGO Stage IA1 with lymph-vascular space involvement or stage IA2-IB2).
* Consented for a radical trachelectomy (vaginal/abdominal) or radical hysterectomy (laparoscopic/abdominal).
* Have not started or completed childbearing.
* Strong desire to preserve fertility (trachelectomy group only).
* At least 18 years of age and not older than 45 years at the time of treatment.
* Able to read/ speak the English language.
* Able to provide informed conse

Exclusion Criteria:

* Inability to participate in an informed consent process.
* Patients with a psychiatric disorder precluding response to the survey.
* Patients that are upstaged at the time of surgery and will require adjuvant therapy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with early stage cervical cancer undergoing either radical trachelectomy or radical hysterectomy
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2004-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Assess emotional, sexual and quality of life of women with early stage cervical cancer undergoing radical trachelectomy and to compare same between women undergoing radical trachelectomy versus standard radical hysterectomy (all forms). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Carter, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskcc.org